CLINICAL TRIAL: NCT07265492
Title: UDOPAL Study: Hospital-at-Home Interventional Approach to Pain Management in Patients Receiving Home-Based Hospital Care
Brief Title: UDOPAL Study: Home-Based Interventional Approach to Pain Management in Home-Hospitalized Patients
Acronym: UDOPAL
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital de Manises (Other)
Responsible Party: Principal Investigator, Estefania Romero Serrano, MD, PhD, Principal Investigator, UDOPAL Intervention Program, Pain Medicine Unit, Hospital de Manises, Hospital de Manises
Other Study IDs: UDOPAL; CEIm La Fe Acta N.600-08.10.25 (Registry Identifier: Comité de Ética de la Investigación con medicamentos del CEIM - HOSPITAL UNIVERSITARIO Y POLITÉCNICO LA FE)
Record Dates: First submitted 2025-11-17; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain; Cancer Pain; Neuropathic Pain; Palliative Care
Keywords: UDOPAL; Home Hospitalization; Palliative Care; Palliative Pain Care; Nerve Blocks; Chronic Pain; Cancer Pain; Pain Relief; Opioid Reduction; Multidisciplinary Model; Hospital-at-Home; Home Health Care; Home Medical Services; Integrated Home Care; Hospital in the Home; Domiciliary Care; Home-Based Hospital Care; Interventional Pain Management
MeSH Terms: conditions — Chronic Pain; Cancer Pain; Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UDOPAL Cohort Description: Prospective observational cohort including patients admitted
  Interventions: Other: UDOPAL model

INTERVENTIONS:
Other: UDOPAL model — The UDOPAL model proposes a novel clinical approach to manage pain in patients hospitalized at home through the use of interventional pain techniques.
  The model enables trained home-hospitalization professionals to perform minimally invasive, ultrasound-guided procedures at the patient's home when conventional pharmacological strategies are insufficient.
  This observational study evaluates the feasibility, safety, and clinical effectiveness of this innovative home-based pain management approach, focusing on pain intensity reduction, opioid-sparing effect, improvement in functional status, and patient and family satisfaction.

SUMMARY:
The UDOPAL Study proposes an innovative home-based care approach for the management of pain in patients admitted to the Home Hospitalization Unit (UHD). This model incorporates interventional pain management techniques into the clinical practice of home-hospital professionals, supported when necessary by specialists from the Pain Medicine Unit.

Pain is a prevalent and often undertreated problem in patients receiving home hospitalization, where complex or oncologic pain may require specialized procedures that traditionally are only performed in hospital settings. The UDOPAL model aims to bridge this gap by providing ultrasound-guided and minimally invasive pain procedures directly at the patient's home, including nerve blocks, infiltrations, and other targeted interventions.

This observational, prospective study evaluates the feasibility, safety, and clinical impact of implementing interventional pain management at home. Adult patients with chronic, oncologic, or complex pain will be included. Outcomes include pain intensity, opioid use, functional improvement, quality of life, and patient satisfaction, as well as adverse events related to the techniques.

The study seeks to provide scientific evidence supporting a new model of interventional home-based pain care that improves comfort, continuity of care, and efficient use of healthcare resources. The project was approved by the Ethics Committee (CEIm Hospital Universitario y Politécnico La Fe, Acta No. 600, 08/10/2025) and is conducted at Hospital de Manises (Valencia, Spain).

DETAILED DESCRIPTION:
Introduction

Pain is one of the most prevalent and distressing symptoms among patients receiving home hospitalization, especially those with chronic or oncologic conditions. Despite the advances in home-based medicine, the management of moderate to severe pain continues to be a clinical challenge. Conventional pharmacological treatment alone is often insufficient, and access to specialized interventional pain techniques remains limited to hospital settings.

In traditional care models, patients experiencing uncontrolled pain must be transferred to the hospital for evaluation or intervention, leading to fragmentation of care, increased healthcare costs, and a significant emotional burden for patients and families. These transfers often disrupt the continuity of palliative and supportive care that the home-hospitalization environment seeks to provide.

The UDOPAL Study (from Unidad del Dolor + Hospitalización Domiciliaria) was designed to address this gap by introducing a structured, collaborative model that enables interventional pain management to be performed safely and effectively at home. This initiative positions home-hospital professionals at the center of the intervention, empowering them to deliver advanced pain procedures within the patient's own environment, supported by the Pain Medicine Unit when required.

The study reflects an evolution in the concept of pain management-shifting from a hospital-centered model to an integrated, patient-centered continuum of care. The UDOPAL model aligns with the principles of the World Health Organization and modern palliative medicine, emphasizing early, multidisciplinary, and accessible interventions that improve comfort, dignity, and quality of life.

Beyond clinical innovation, the UDOPAL project also represents an organizational and educational advance: it introduces a systematic training framework for home-hospital professionals to perform ultrasound-guided and minimally invasive procedures for pain control, under a protocolized supervision system. This dual focus-clinical and educational-aims to ensure safety, reproducibility, and scalability of the model.

Objectives and Hypothesis

The UDOPAL Study is based on the hypothesis that interventional pain management procedures-when adapted, standardized, and safely performed by trained Home Hospitalization Unit (UHD) professionals-can improve pain control, functionality, and patient satisfaction while optimizing healthcare resource utilization.

Primary Objective

To evaluate the feasibility and safety of performing interventional pain management techniques at home by UHD professionals within the UDOPAL model.

Secondary Objectives

To describe the prevalence and intensity of pain among patients admitted to a Home Hospitalization Unit and to determine the proportion experiencing mild, moderate, or severe pain.

To measure the reduction in opioid consumption, assessing whether improved pain control leads to decreased opioid requirements and fewer adverse effects.

To analyze the improvement in patient functionality, evaluating whether better pain management reduces physical limitations and enhances functional capacity.

To assess whether the UDOPAL model contributes to an increase in patients' quality of life.

To evaluate patient and family satisfaction with pain management and overall home-based care.

To explore the professional perception of the model's clinical impact among UHD and Pain Unit staff.

To assess the implementation of the UDOPAL model in real clinical practice, identifying facilitators and barriers to its adoption.

To analyze the healthcare demand generated by the UDOPAL model, including its influence on workload, care coordination, and service utilization.

The working hypothesis is that the UDOPAL model will demonstrate high feasibility, a favorable safety profile, and significant clinical and organizational benefits compared to conventional home-based care, contributing to a more integrated, efficient, and patient-centered approach to pain management at home.

Study Design

The UDOPAL Study is an observational, prospective study designed to evaluate the early implementation of a novel home-based model for pain management in patients admitted to the Home Hospitalization Unit (UHD). The model integrates interventional pain procedures into standard clinical practice at home, performed by UHD professionals trained in the UDOPAL protocol, with support from the Pain Medicine Unit.

The study assesses the impact of this integrated model on clinical, organizational, and perceived-quality outcomes, comparing results obtained before and after the implementation of the UDOPAL protocol. Particular attention is given to the effects of early intervention during the initial stages of clinical complexity, when timely pain control may influence the overall course of illness and quality of life.

Study Population

Adult patients (≥18 years) admitted to the Home Hospitalization Unit who present acute, chronic, or oncologic pain and may benefit from interventional pain procedures. Patients are identified by UHD professionals and managed according to the UDOPAL protocol once the intervention phase begins.

Inclusion Criteria

Patients admitted to the UHD.

Presence of acute, chronic, or oncologic pain requiring advanced pain management.

Indication for interventional pain techniques (e.g., peripheral nerve blocks, infiltrations, pulsed radiofrequency).

Ability to understand and sign informed consent (or through a legal representative).

Exclusion Criteria

Contraindication to interventional techniques (coagulopathy, local infection, allergy to local anesthetics).

Cognitive impairment or communication barrier that prevents adequate assessment.

Absence of safe or logistically feasible home environment.

Intervention and Comparison

The UDOPAL model is implemented as an early intervention protocol combining pharmacologic optimization with minimally invasive pain procedures performed at the patient's home. UHD professionals trained under the UDOPAL framework conduct the interventions using portable ultrasound guidance and aseptic technique.

The study compares two periods:

Pre-intervention phase: standard home-hospitalization care before UDOPAL implementation.

Post-intervention phase: care delivered under the UDOPAL protocol, integrating interventional pain management.

Variables and Data Collection

Clinical and service indicators are prospectively collected and compared between phases, including:

Pain intensity (VAS/NRS).

Opioid consumption (morphine-equivalent daily dose).

Functional capacity and mobility.

Quality of life and satisfaction of patients and families.

Professional perception of impact on care quality.

Resource utilization: emergency visits, hospital readmissions, and assistance demand.

Sample Size and Duration

Approximately 80-100 patients are expected to be included during a 12-month recruitment period. The sample size is pragmatic, based on UHD patient flow and expected feasibility of early intervention.

Statistical Analysis

Descriptive statistics will be used for baseline characteristics. Continuous variables will be compared between pre- and post-intervention phases using paired t-test or Wilcoxon signed-rank test, as appropriate. Categorical variables will be compared using χ² or Fisher's exact test. A p-value <0.05 will be considered statistically significant.

Ethical Considerations

The study was approved by the Ethics Committee (CEIm Hospital Universitario y Politécnico La Fe, Acta No. 600, 08/10/2025). Written informed consent will be obtained from all participants. The study follows the Declaration of Helsinki and Good Clinical Practice guidelines.

Implementation and Training Framework

The UDOPAL Study is both a clinical and educational initiative aimed at ensuring that interventional pain techniques can be safely and effectively performed within the home-hospitalization environment. The model is implemented through structured professional training, standardized clinical protocols, and continuous quality evaluation.

Professional Training

Before implementation, UHD professionals (physicians and nurses) participate in a dedicated educational program coordinated by the Pain Medicine Unit. The curriculum combines theoretical modules-covering pain pathophysiology, pharmacologic optimization, and indications for interventional techniques-with practical ultrasound-guided workshops. Training emphasizes aseptic technique, patient selection, prevention of complications, and post-procedure follow-up.

Clinical Implementation

After completing training, UHD professionals progressively incorporate interventional pain procedures into their clinical practice, following the standardized UDOPAL protocol. Pain specialists from the Pain Medicine Unit remain available for consultation and case review, ensuring adherence to safety standards and technical consistency.

Safety and Quality Assurance

Safety is continuously monitored through the recording of procedure-related complications, unplanned hospital visits, and any adverse events. A predefined escalation pathway allows for immediate hospital transfer if necessary. All data are documented in a secure electronic case report form and reviewed monthly by the UDOPAL coordination team.

Implementation Assessment

The implementation process is evaluated using both quantitative and qualitative indicators:

Quantitative indicators: number and type of procedures performed, success rate, complication rate, and time to pain relief.

Qualitative indicators: professional perception of feasibility, coordination between units, and satisfaction with the training received.

Expected Impact and Conclusions

The UDOPAL Study seeks to generate clinical evidence supporting the feasibility and safety of performing interventional pain procedures within the home-hospitalization setting. By incorporating these techniques into early stages of patient management, the model aims to achieve more effective pain control, reduce opioid requirements, and improve functional capacity and perceived quality of life.

In addition to its direct clinical benefits, the project is expected to strengthen collaboration between the Home Hospitalization Unit and the Pain Medicine Unit, promoting shared decision-making and continuity of care. The implementation process will also provide valuable insight into the practical challenges of integrating interventional pain management into routine domiciliary care.

The results of this study will help define safe practice standards for interventional pain techniques performed at home and may inform future guidelines for comprehensive pain management in home-based patients.

The UDOPAL Study represents a step toward more personalized, multidisciplinary, and accessible care for patients experiencing pain during home hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) admitted to the Home Hospitalization Unit (UHD) of the Manises Health Department.
* Presence of active pain, classified as mild, moderate, or severe.
* Clinical assessment indicating suitability for interventional pain management, as determined by a UDOPAL-trained physician.
* Physical and clinical conditions that allow the performance of interventional procedures at home under standardized safety precautions.
* Signed informed consent obtained from the patient and/or a legally authorized representative in cases of incapacity.

Exclusion Criteria:

* Very limited life expectancy (estimated survival <72 hours) or terminal/agonal condition.
* Contraindication to interventional pain procedures, including:

  1. Uncorrectable coagulopathy.
  2. Systemic infection or local infection at the puncture site.
  3. Documented allergy to any of the planned medications.
  4. Tumor located in the infiltration area.
  5. Pregnancy or breastfeeding.
* Altered level of consciousness or severe cognitive impairment without a responsible family member or without the possibility of obtaining valid informed consent.
* Home environment conditions that do not ensure minimal hygiene, safety, or logistical support (e.g., inadequate lighting, lack of privacy, insufficient family assistance, or limited access for the medical team).
* Explicit refusal by the patient and/or family to undergo interventional pain procedures.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Home Hospitalization Unit (HHU) of the Manises Health Department who present with acute, chronic, oncologic, or complex pain requiring assessment for interventional pain management at home. The study population includes individuals with adequate clinical stability to undergo minimally invasive procedures in the domiciliary setting, as evaluated by a UDOPAL-trained physician. Patients may present a wide range of pain etiologies, functional limitations, or palliative needs commonly managed during home hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-08 (Estimated); Study Completion 2026-10-08 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Intensity (Numeric Rating Scale, NRS 0-10) | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Pain intensity will be assessed using the Numeric Rating Scale (NRS, 0-10) for patients able to self-report pain.
  The primary outcome represents the mean reduction in NRS pain intensity from baseline to each follow-up point.
Change in Pain Intensity (PAINAD 0-10 for patients with cognitive impairment) | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Pain intensity will be assessed using the Pain Assessment in Advanced Dementia Scale (PAINAD, 0-10) for patients with cognitive impairment or communication difficulties.
  The primary outcome represents the mean reduction in PAINAD score from baseline to each follow-up point.

SECONDARY OUTCOMES:
Opioid Consumption | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Daily opioid use will be converted into oral morphine equivalent dose (mg/day) and compared across all follow-up points. The outcome evaluates the potential opioid-sparing effect of home-based interventional pain management.
Functional Status | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Functional capacity will be measured using the Barthel Index (0-100), comparing baseline scores with those at 1 week, 1 month, and at discharge.
Patient and Family Satisfaction | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Satisfaction with pain control and overall home-based care will be assessed using a 5-point Likert scale questionnaire at discharge and 1 month.
Professional Perception of Feasibility | baseline and at completion of the implementation phase (approximately 1 month)
  UHD professionals will complete a structured survey on the perceived feasibility, safety, and impact of interventional pain management at home after the first implementation phase.
Change in Quality of Life (EQ-5D-5L Score) | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Quality of life will be assessed using the EuroQOL-5D-5L (EQ-5D-5L) questionnaire, which measures mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  The outcome represents the change in the EQ-5D-5L index score and visual analogue scale (VAS) between baseline and follow-up time points to evaluate the patient's perceived health status during home hospitalization.
Change in Functional Status (Barthel Index) | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Functional capacity will be assessed using the Barthel Index (0-100), which measures performance in activities of daily living (ADL), including feeding, bathing, mobility, and continence.
  The outcome represents the change in total Barthel Index score between baseline and follow-up time points to evaluate improvement in autonomy and physical function after home-based interventional pain management.
Change in Analgesic Consumption Profile | Baseline (Day 0), 24 hours, 48 hours, 1 week, 1 month, and at discharge from the Home Hospitalization Unit (HHU)
  Analgesic treatment will be recorded and classified into the following categories:
  Opioids: converted to daily oral morphine equivalent dose (mg/day, DEM).
  Adjuvant Analgesics: antidepressants, anticonvulsants, or other neuromodulators.
  Corticosteroid Adjuvants: such as dexamethasone or equivalents.
  Non-opioid Analgesics: acetaminophen and/or nonsteroidal anti-inflammatory drugs (NSAIDs).
  The outcome represents the change in analgesic use across all categories between baseline and follow-up assessments, to evaluate potential opioid-sparing effects and optimization of multimodal analgesia after implementation of home-based interventional pain management.
Incidence of Adverse Events Related to Home-Based Interventional Pain Procedures | From procedure initiation until 1 month follow-up or discharge from the Home Hospitalization Unit (HHU), whichever occurs later
  All adverse events occurring during or after interventional pain procedures performed at home will be prospectively recorded.
  Events will be categorized as:
  Immediate procedural events: e.g., local bleeding, vasovagal reaction, accidental puncture, or transient nerve irritation.
  Delayed complications: e.g., infection, hematoma, increased pain, or unexpected neurological symptoms.
  Systemic or medication-related events: e.g., allergic reaction, sedation, nausea, or cardiovascular changes associated with local anesthetics or corticosteroids.
  Each event will be graded according to its severity (mild, moderate, severe) and its relationship to the procedure (related, possibly related, unrelated).
Rate of Unplanned Hospital Transfers | From procedure initiation until 1 month follow-up or discharge from the Home Hospitalization Unit , whichever occurs later
  The outcome measures the proportion of patients who required unplanned transfer or readmission to the hospital during or after home-based interventional pain management.
  Transfers may result from uncontrolled pain, procedure-related complications, or other medical reasons. Each event will be documented with its cause, timing, and relationship to the home-based procedure.
  This indicator reflects the safety and feasibility of maintaining patients under home-hospitalization care while receiving interventional pain management.
Number of Interconsultations Between the Home Hospitalization Unit and the Pain MedicineUnit | Throughout the entire home-hospitalization episode and during the 1-month follow-up period
  The outcome measures the total number of interconsultations or collaborative case discussions between UHD professionals and the Pain Medicine team related to home-based pain management procedures.
  Each interconsultation will be recorded prospectively, specifying its reason (e.g., indication for interventional technique, pharmacologic adjustment, follow-up review), mode of communication (in-person, phone, or telematic), and outcome of the consultation.
  This indicator reflects the level of interdisciplinary collaboration and coordination required to sustain the home-based interventional pain management model.
Response Time From Indication to Procedure Completion | From clinical indication to completion of the interventional procedure (measured for each patient during the home-hospitalization episode)
  The outcome measures the elapsed time between the clinical indication for a home-based interventional pain procedure and its actual performance by the UHD team.
  The interval (in hours) will be recorded for each case, starting from the documented medical indication to the completion of the procedure.
  This indicator evaluates the responsiveness and operational efficiency of the UDOPAL model within home-hospitalization care, reflecting how rapidly patients receive interventional pain management once the need is identified.
Total Consultation Time Including Procedure Duration | At each home visit in which an interventional pain procedure is performed
  The outcome measures the total time (in minutes) spent per patient visit when an interventional pain technique is performed at home.
  The measurement includes the complete duration of the home consultation-from the start of patient assessment to the end of the interventional procedure-and accounts for preparation, execution, and immediate post-procedure monitoring.
  This indicator evaluates the time investment required for each intervention and contributes to assessing the overall efficiency and workload associated with home-based interventional pain management.
Number of Interventional Pain Procedures Performed at Home | tecniques per patient/ tecniques per month
  The outcome measures the total number and type of interventional pain management procedures performed at the patient's home by UHD professionals.
  Each procedure will be prospectively recorded, specifying the anatomical region, technique used (e.g., peripheral nerve block, trigger point infiltration, paravertebral block), medications administered, and whether the procedure was completed successfully.
  This indicator reflects the clinical activity, feasibility, and procedural performance of home-based interventional pain management within the UDOPAL model.
Number of Patients Undergoing Interventional Pain Procedures at Home | tecniques per patient
  The outcome measures the total number and proportion of patients who receive one or more interventional pain management techniques during their home-hospitalization episode.
  For each patient, the type and number of procedures performed will be documented, including peripheral nerve blocks, infiltrations, or other ultrasound-guided techniques.
  This indicator reflects the clinical applicability and penetration of home-based interventional pain management within the UDOPAL model.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared outside the research team. The dataset contains sensitive clinical information from home-hospitalized patients, and data sharing is not included in the current ethics approval or informed consent.